CLINICAL TRIAL: NCT02222064
Title: Exploratory Study of Mindfulness for Inpatients With Chronic Gastrointestinal Pain: Does it Reduce Pain Related Distress and Increase Confidence in Pain Self-management?
Brief Title: Pilot of Mindfulness Therapy for Inpatients With Gastro-intestinal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14/0190
Record Dates: First submitted 2014-08-12; First posted 2014-08-21 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-05

CONDITIONS: Gastro-intestinal Pain
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness (Experimental): 8 week self-managed mindfulness based intervention
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness is a psychological intervention based on increasing skills of non-judgemental awareness using meditations. In this study a self-directed 8 week course of mindfulness will be used involving self-help materials in the form of a book and 8 guided meditations on audio files.

SUMMARY:
Research questions/hypotheses

1. Can an individual mindfulness intervention for Gastro Intestinal Failure inpatients reduce pain-related distress, improve quality of life, and increase confidence in pain self-management?
2. How useful and applicable do Gastro Intestinal Failure inpatients find Mindfulness methods?

ELIGIBILITY:
Inclusion Criteria:

* >18 years, pain experienced
* >3 months, proficiency in English

Exclusion Criteria:

* previous mindfulness experience
* severe cognitive impairment
* profound hearing difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in pain distress rating on 11 point numerical rating scale | Baseline, week 1, week 2, week 3, week 4, week 5 , week 6, week 7, week 8
  A numerical rating scale scored from 0 to 10 which asks "how distressing is the pain on average in the last week with 0 being not distressing at all and 10 being extreme distress"

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | At baseline, week 8
Pain Self Efficacy Questionnaire | At baseline, week 8
  a 10 item scale that attempts to capture a measure of individual's confidence in being active despite pain, rated on a numerical scale from 0 "not at all confident" to 6 "completely confident"
Chronic Pain Acceptance Questionnaire | At baseline, week 8
  a 20 item measure included to provide a rating of acceptance of pain
Five Facet Mindfulness Questionnaire | At baseline, week 8
  a 39 item questionnaire which has been developed from five mindfulness questionnaires using exploratory factor analysis
Self-report record of using mindfulness exercises (frequency and duration) | Week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8
Brief account of experience of pain and doing the mindfulness exercises | Week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8
  participants will be asked to write a brief (<1 page) account of their experience of their pain and of doing the mindfulness exercises over the preceding week
Change in pain intensity rating on 11 point numerical rating scale | Baseline, week 1, week 2, week 3, week 4, week 5 , week 6, week 7, week 8
  A numerical rating scale scored from 0 to 10 which asks "how intense is the pain on average in the last week with 0 being no pain and 10 being extreme pain"

CONTACTS AND LOCATIONS:
Locations (1):
- University College Hospital, London, United Kingdom